CLINICAL TRIAL: NCT06504446
Title: A Phase 2b, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy, Safety, and Tolerability of Taplucainium Inhalation Powder (NOC-110) in Adults With Refractory or Unexplained Chronic Cough
Brief Title: Study to Assess the Efficacy, Safety, and Tolerability of NOC-110 in Adults With Refractory or Unexplained Chronic Cough
Acronym: ASPIRE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nocion Therapeutics (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NOC110-C-202
Record Dates: First submitted 2024-07-11; First posted 2024-07-16 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Refractory or Unexplained Chronic Cough

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- NOC-110 1mg (Experimental): NOC-110 (taplucainium) administered by daily dry powder inhalation. NOC-110 contains a dry powder lactose blend containing drug substance taplucainium administered using an available inhaler.
  Interventions: Drug: NOC-110
- NOC-110 3mg (Experimental): NOC-110 (taplucainium) administered by daily dry powder inhalation. NOC-110 contains a dry powder lactose blend containing drug substance taplucainium administered using an available inhaler.
  Interventions: Drug: NOC-110
- NOC-110 6mg (Experimental): NOC-110 (taplucainium) administered by daily dry powder inhalation. NOC-110 contains a dry powder lactose blend containing drug substance taplucainium administered using an available inhaler.
  Interventions: Drug: NOC-110
- Placebo (Placebo Comparator): The matching placebo contains inhalation grade lactose blended with arginine. The blend is taste masked to the active drug product to minimize unblinding due to taste differences.
  The matching placebo will be administered via the same inhaler.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: NOC-110 — Inhalation powder
  Other Names: taplucainium
  Arms: NOC-110 1mg; NOC-110 3mg; NOC-110 6mg
Other: Placebo — Inhalation powder
  Arms: Placebo

SUMMARY:
This is a phase 2b, randomized, double-blind, placebo-controlled study investigating the efficacy, safety, and tolerability of Taplucainium Inhalation Powder (NOC-110) once daily in adults with refractory or unexplained chronic cough.

DETAILED DESCRIPTION:
Approximately 455 participants will take part in the study. It is anticipated that up to 1264 participants will be screened. Participation will be approximately 13 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Refractory or unexplained chronic cough for ≥ 12 months.
* Women of childbearing potential agree to follow the protocol specified contraceptive - guidance during the study.
* Males who are not vasectomized must agree to use the contraceptive methods defined in the protocol.
* Able to provide Informed Consent.

Exclusion Criteria:

* Previous exposure to taplucainium (formerly NTX-1175) or known allergy or hypersensitivity to taplucainium, its excipients/metabolites, or related compounds.
* Participants who are currently participating in another drug or device clinical study
* Participants who have participated in an Acute or Chronic Cough investigational study within 60 days before the start of the Screening.
* Current diagnosis of chronic obstructive pulmonary disease, bronchiectasis, unexplained pulmonary fibrosis, hemoptysis, bronchial asthma, or other pulmonary disease.
* Respiratory tract infection within 4 weeks of Screening or during screening period.
* Any female who is pregnant or lactating or wishing to become pregnant.
* Donation of > 1 Unit (450 milliliter or more) of blood within 60 days prior to the first dosing.
* Alcohol or drug use disorder within the past 2 years.
* Current smoker/vaper or individuals who have given up smoking within the past 6 months of screening, and/or those with >20 pack-year smoking history.
* Current opiate/opioid use or medical history of opiate/opioid use disorder.
* History of concurrent malignancy or recurrence of malignancy in the last 2 years.
* Body Mass Index of ≥40 kg/m2.
* Positive results for human immunodeficiency virus, hepatitis B, or hepatitis C virus.
* Unable to refrain from the use of medications and treatments that can impact cough during the study.
* Have clinically significant history or evidence of poorly controlled cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, neurological, immunological, or psychiatric disorder(s).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 455 (Estimated)
Dates: Start 2024-09-24 (Actual); Primary Completion 2026-04-10 (Estimated); Study Completion 2026-04-10 (Estimated)

PRIMARY OUTCOMES:
Change in 24-hour Coughs per hour from Baseline | Baseline to End of Treatment
  Change in 24-hour Coughs per hour from Baseline will be based on VitaloJAK® Cough Counts. The VitaloJAK® is a 510(k)-cleared medical device consisting of a digital sound recorder with 2 microphones; a lapel air microphone attached to the participant's clothing and an adhesive chest wall microphone which is attached to the skin at the top of the sternum.

SECONDARY OUTCOMES:
Change in Awake coughs per hour from Baseline | Baseline to End of Treatment
  Change in Awake coughs per hour from Baseline will be based on VitaloJAK® Cough Counts. The VitaloJAK® is a 510(k)-cleared medical device consisting of a digital sound recorder with 2 microphones; a lapel air microphone attached to the participant's clothing and an adhesive chest wall microphone which is attached to the skin at the top of the sternum.
Change in the Cough Severity Visual Analog Scale from Baseline | Baseline to End of Treatment
  Visual Analogue Scales for Cough Severity (CS-VAS) will be performed as outlined in the Schedule of Assessments. Participants rate the severity of their cough by marking on the horizontal line their cough severity, with the extreme left side of the line represents "no cough" and the extreme right side of the line representing "worst cough."
Change in the Urge to Cough Visual Analog Scale from Baseline | Baseline to End of Treatment
  Urge to Cough Analogue Scales for Cough Severity (UC-VAS) will be performed as outlined in the Schedule of Assessments. Participants rate the severity of their cough by marking on the horizontal line their cough severity, with the extreme left side of the line represents "no cough" and the extreme right side of the line representing "worst cough."
Change in the Leicester Cough Questionnaire from Baseline | Baseline to End of Treatment
  Leicester Cough Questionnaire (LCQ) is a validated cough-specific quality of life measure that evaluates the impact of cough across 3 domains: physical, psychological, and social. The LCQ is a 19-item questionnaire with each item scored using a 7-point Likert scale ranging from 1 = all the time to 7=none of the time. The total severity score ranges from 3-21, with a lower score indicating greater impairment of health status due to cough.
Patient Global Impressions of Improvement score | End of Treatment
  Patient Global Impressions of Improvement (PGI-I) is used to assess improvement or worsening of the Participants status in relation to the therapeutic area of interest. The main purpose of the scale is to quantify the extent to which the participant has improved or deteriorated over time. The PGI-I is a 7-point Likert scale ranging from 1=Very Much Better to 7=Very Much Worse.
Incidence and severity of adverse events and serious adverse events | Baseline to End of Treatment

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Frankel, MD, Study Director — Chief Medical Officer Nocion Therapeutics, Inc.
Locations (106):
- United States (68):
  - G & L Research, LLC, Foley, Alabama
  - Medical Research of Arizona, Scottsdale, Arizona
  - AMR Phoenix, Tempe, Arizona
  - Little Rock Allergy & Asthma, P.A. Clinical Research Center, Little Rock, Arkansas
  - So Cal Clinical Research, Huntington Beach, California
  - Allergy and Asthma Associates of Southern California dba Southern California Research, Laguna Niguel, California
  - Paradigm Clinical Research Centers, LLC - Modesto, Modesto, California
  - NewportNativeMD,Inc, Newport Beach, California
  - Center for Clinical Trials, LLC, Paramount, California
  - Paradigm Clinical Research Centers, LLC, Redding, California
  - DaVinci Research LLC., Roseville, California
  - Allergy & Asthma Associates of Santa Clara Valley, San Jose, California
  - California Allergy & Asthma Medical Group Inc., San Jose, California
  - Allergy, Asthma, and Immunology Medical Group, Ventura, California
  - Allergy and Asthma Clinical Research Inc, Walnut Creek, California
  - Lynn Institute of Denver, Aurora, Colorado
  - Innovative Research of West Florida, Inc., Clearwater, Florida
  - Omega Research Debary, LLC, DeBary, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Clinical Site Partners, LLC Leesburg dba Flourish Research, Leesburg, Florida
  - Suncoast Research Group, LLC Miami - Little Havana dba Flourish Research, Miami, Florida
  - Well Pharma Medical Research Corporation, Miami, Florida
  - University of South Florida - PARENT, Tampa, Florida
  - Clinical Site Partners, LLC Orlando dba Flourish Research, Winter Park, Florida
  - Aeroallergy Research Laboratories of Savannah, Inc., Savannah, Georgia
  - Duly Health and Care, Winfield, Illinois
  - Accellacare of McFarland Clinic, Ames, Iowa
  - The Iowa Clinic, PC, West Des Moines, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Bluegrass Allergy Research, Lexington, Kentucky
  - Allergy & Asthma Specialists, PSC, Owensboro, Kentucky
  - Continental Clinical Solutions, LLC, Towson, Maryland
  - Infinity Medical Research Inc, Russells Mills, Massachusetts
  - Clinical Research Institute, Minneapolis, Minnesota
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - The Curators of the University of Missouri on behalf of University of Missouri Health Care, Columbia, Missouri
  - Midwest Chest Consultants, Saint Charles, Missouri
  - Sundance Clinical Research, St Louis, Missouri
  - The Clinical Research Center, LLC, St Louis, Missouri
  - Montana Medical Research, Inc., Missoula, Montana
  - AMR Las Vegas, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Allergy Partners of New Jersey P C, Ocean City, New Jersey
  - The Valley Hospital, Paramus, New Jersey
  - St Josephs Physicians Med PC Pulmonary Health, Liverpool, New York
  - Equity Medical LLC, New York, New York
  - Allergy Partners Clinical Research, Asheville, North Carolina
  - Clinical Research of Gastonia, Gastonia, North Carolina
  - M3 Wake Research, Inc., Raleigh, North Carolina
  - Accellacare, Winston-Salem, North Carolina
  - Southeastern Research Center LLC, Winston-Salem, North Carolina
  - Remington-Davis, Inc., Columbus, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Vital Prospects Clinical Research Institute, P.C., Tulsa, Oklahoma
  - Northwest Research Center, Portland, Oregon
  - Suburban Research Associates, West Chester, Pennsylvania
  - Care Access Research - Warwick 1, Warwick, Rhode Island
  - Lowcountry Lung and Critical Care, P.A., Charleston, South Carolina
  - Accellacare, Mt. Pleasant, South Carolina
  - Clinical Research of Rock Hill, Rock Hill, South Carolina
  - Internal Medicine and Pediatric Associates of Bristol, PC, Bristol, Tennessee
  - Accellacare d/b/a Accellacare of Knoxville, Knoxville, Tennessee
  - Pharmaceutical Research & Consulting, Inc., Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - South Texas Allergy & Asthma Medical Professionals, San Antonio, Texas
  - Alamo ENT Associates, San Antonio, Texas
  - TPMG Clinical Research Williamsburg, Williamsburg, Virginia
  - Allergy, Asthma & Sinus Center, SC, Greenfield, Wisconsin
- Belgium (4):
  - UZ Leuven, Leuven
  - AZ Sint-Maarten, Mechelen
  - Pneumocare, Namur
  - AZ Delta, Roeselare
- Canada (10):
  - Dynamic Drug Advancement, Ajax, Ontario
  - BLC Clinical Research, Burlington, Ontario
  - McMaster University, Hamilton, Ontario
  - Inspiration Research Limited, Toronto, Ontario
  - Recherche GCP Research, Montreal, Quebec
  - DIEX Recherche Quebec Inc., Québec, Quebec
  - Clinique Specialisee en Allergie de la Capitale, Québec, Quebec
  - Clinique de pneumologie et du sommeil de Lanaudière, Saint-Charles-Borromée, Quebec
  - DIEX Recherche Sherbrooke Inc., Sherbrooke, Quebec
  - DIEX Recherche Victoriaville Inc., Victoriaville, Quebec
- Germany (8):
  - Pneumologisches Studienzentrum Muenchen West, Munich, Bavaria
  - Lungenzentrum Darmstadt, Darmstadt, Hesse
  - Medaimun GmbH, Frankfurt am Main, Hesse
  - Zentrum fuer ambulante pneumologische Forschung Marburg GbR, Marburg, Hesse
  - Pneumologicum Halle, Halle, Saxony-Anhalt
  - Pneumologisches Forschungsinstitut Hohegeest GbR, Geesthacht, Schleswig-Holstein
  - Velocity Research Germany GmbH, Lübeck, Schleswig-Holstein
  - Pneumologisches Studienzentrum MVZ "Die Lungenärzte", Berlin, State of Berlin
- Poland (8):
  - Prywatny Gabinet Internistyczno-Alergologiczny, Bialystok
  - Prywatna Praktyka Lekarska Gabinet Pediatryczno-Alergologiczny, Bialystok
  - Centrum Medyczne Pratia Bydgoszcz, Bydgoszcz
  - Centrum Medyczne Pratia Czestochowa, Częstochowa
  - Ostrowieckie Centrum Medyczne spółka cywilna Anna Olech-Cudzik, Krzysztof Cudzik, Ostrowiec Świętokrzyski
  - Centrum Medyczne Lucyna Andrzej Dymek s.c., Strzelce Opolskie
  - Gabinet Pulmonologii i Diagnostyki Chorób Alergicznych Dorota Maria Małosek, Szczecin
  - Alergo-Med Specjalistyczna Przychodnia Lekarska Sp. Z .O.O., Tarnów
- United Kingdom (8):
  - Ormeau Clinical Trials Ltd, Belfast, Belfast
  - Belfast City Hospital, Belfast, Belfast
  - West Walk Surgery, Bristol, Bristol
  - Castle Hill Hospital, Cottingham, East Riding of Yorkshire
  - King's College Hospital, London, Greater London
  - Wythenshawe Hospital, Wythenshawe, Greater Manchester
  - Nottingham City Hospital, Nottingham, Nottinghamshire
  - North Tyneside General Hospital, North Shields, Tyne & Wear